CLINICAL TRIAL: NCT03175458
Title: Schnederian Membrane Elevation and Augmentation With Deproteinized Bovine Bone [Tutu-gen Bone] Versus Graft Less Tenting Technique With Simultaneous Implant Placement: Randomized Clinical Trial
Brief Title: Schnederian Membrane Elevation and Augmentation With Deproteinized Bovine Bone [Tutu-gen Bone] Versus Graft Less Tenting Technique With Simultaneous Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed Fouad Mahmoud, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cebc.cu
Record Dates: First submitted 2017-05-17; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Maxillary Sinus Floor Elevation
Keywords: tenting; grafting; implant placement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sinus lift,implant placement,tenting (Experimental): elevation of the sinus membrane with simultaneous implant placement without the use of any bone graft material(tenting technique)
  Interventions: Procedure: sinus lift,implant placement,tenting
- sinus lift,implant placement,bovine bone (Active Comparator): elevation of the sinus membrane with simultaneous implant placement together with deproteinized bovine bone graft substitute for augmentation
  Interventions: Procedure: sinus lift,implant placement,bovine bone

INTERVENTIONS:
Procedure: sinus lift,implant placement,tenting — elevation of the sinus membrane then insertion of the implants without any bone graft material( graft-less) for augmentation
  Arms: sinus lift,implant placement,tenting
Procedure: sinus lift,implant placement,bovine bone — sinus membrane elevation then placement of the implants together with deproteinized bovine bone substitute as a graft material for augmentation
  Arms: sinus lift,implant placement,bovine bone

SUMMARY:
30 recruited patients indicated for sinus membrane elevation with simultaneous implant placement. patients are divided into 2 groups each group contain 15 patients, one group assigned for placement of bovine bone graft after membrane elevation and insertion of the implants while the other group assigned for graft-less tenting technique after membrane elevation and insertion of the implant.

DETAILED DESCRIPTION:
On the 2 groups a mucoperiosteal flap is elvated then a lateral wondow is created then sinus membrane is elevated then the implants are placed, in the control group deproteinized bovine bone graft substitute is placed in the sinus for augmentation while in the study group no bone graft is added inside the sinus( graftless tenting technique)

ELIGIBILITY:
Inclusion Criteria:

* patients with atrophic maxilla and pneumatization of the maxillary sinus with residual bone height at least 5mm as per MISCH criteria.
* both sexes.

Exclusion Criteria:

* sinus pathology
* heavy smokers(more than 20 cigarettes per day.
* patients with systemic disease that may affect normal healing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 7 days post operative
  evaluation of post operative complications in terms of pain and edema using patient pain chart

SECONDARY OUTCOMES:
implant stability | will be measured intraoperatively immediately after insertion of the implants and will be measure one more time 6 months after the 1st operation at the time of exposure of the implants
  measurement of the implant stability using the osstell device
height of bone gained or lost around the implants | 6 months postoperative
  two cone beam computed tomography(CBCT) will be taken for the patient, one immediate postoperative and the other 6 months after the operation then the height of bone gained or lost around the implants will be assessed by superimposing the same section in the two CBCTS.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided